CLINICAL TRIAL: NCT06496685
Title: Dog Assisted Therapy Program for Children With Attention Deficit Hyperactivity Disorder: a Randomized Clinical Trial
Brief Title: Dog Assisted Therapy Program for Children With ADHD
Acronym: DOGAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P18/079
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Animal Assisted Therapy
Keywords: Animal Assisted Therapy; Attention Deficit Disorder with Hyperactivity; Children; Primary Health Care Center; Psychotherapy; Psychiatry
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Participants were recruited from a community Child and Adolescent Mental Health Service and a Primary Health Care Center. And randomized in two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group carried out a total of 14 one-hour group sessions, on a weekly basis for 14 consecutive weeks. The groups were formed by 8 participants. Sessions included the participation of one certified therapy dog, one technician specialized in AAT and a psychologist. Participants received their usual treatment (pharmacological and/or individual and family cognitive-behavioral treatment).
  Intervention:
  All sessions: Establishment of structured routines and schedules to help the child organize and manage daily responsibilities. Positive reinforcement to reward and motivate desirable behaviors.
  Sessions 1-7: Impulsivity management techniques. Social skills training. Self-control techniques to identify and manage moments of impulsivity.
  Sessions 8-14: Reinforcement of attention and concentration through strategies such as dividing tasks into smaller, more manageable parts. Cognitive-behavioral therapy to work on self-esteem, self-control and problem solving.
  Interventions: Other: psychoeducational
- Control Group (No Intervention): Treatment as usual (pharmacological and/or individual and family cognitive-behavioral treatment).

INTERVENTIONS:
Other: psychoeducational — A structured AAT program and usual treatment in Experimental group.
  Other Names: Animal Assisted Therapy
  Arms: Experimental Group

SUMMARY:
The purpose of this study was to evaluate the efficacy of AAT intervention in children with Attention Deficit Hyperactivity Disorder (ADHD), in terms of improving functionality, ADHD-associated symptoms, attention and working memory. Participants were recruited from a community Child and Adolescent Mental Health Service and a Primary Health Care Center. These objectives were accomplished through a multicenter, randomized clinical trial, open-label, two-arm study of AAT for children with ADHD.

DETAILED DESCRIPTION:
The purpose of the present study was to evaluate the efficacy of Animal Assisted Therapy (with therapy dogs) in in children with Attention Deficit Hyperactivity Disorder (ADHD). The investigators conducted a multicenter, randomized, controlled, open-label, two-arm clinical trial. Thirty-six children aged 7-12 diagnosed with ADHD were randomized in two groups. Experimental group: 14 animal assisted therapy (AAT) psychoeducational sessions (once-a-week, 60 minutes) + treatment as usual and control group: treatment as usual. Participants were recruited from a community Child and Adolescent Mental Health Service and a Primary Health Care Center. The investigators evaluated changes on functionality, ADHD-associated symptoms, attention and working memory at pre-treatment and post-treatment. Assessment included intelligence test, ADHD symptoms referred by parents and teacher's (Conners Rating Scale), attention measures (Conners Continuous Performance Test (CPT-3) and children's functioning (Children's Global Assessment Scale (CGAS)).

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 and 12 years old (included).
* Diagnosis of ADHD confirmed at the Child and Adolescent Mental Health Service.
* Intelligence quotient of 80 or higher.
* Delivery of the information sheet and signature of the informed consent.

Exclusion Criteria:

* If in the initial interview they declared having allergy or fear of dogs.
* History of aggression towards animals.
* Co-morbidity with other disorders (conduct disorders, autism spectrum disorders, anxiety disorder or depression).
* If the treatment regimen was modified during the intervention period.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline Children's Global Assessment Scale (CGAS) at 14 weeks. | This scale was administered at baseline and at week 14
  It is a numerical scale to rate the overall functioning of young people under 18 years of age. Scores range from 1 to 100. A higher score indicates better functioning.
Change from baseline Clinical Global Impression - Severity Scale (CGI-S) at 14 weeks | This scale was administered at baseline and at week 14
  Is an instrument for measuring symptom severity of patients with mental disorders. Uses a single item on a Likert scale of seven values from 1= "Normal, not at all ill" to 7= "Among the most extremely ill patients".

SECONDARY OUTCOMES:
Change from baseline Wechsler Intelligence Scale for Children (WISC-IV) at 14 weeks. | This scale was administered at baseline and at week 14
  This instrument measures intellectual ability of children from 6 to 16 years. It was developed to provide an overall measure of general cognitive ability, and measures of intellectual functioning in Verbal Comprehension, Perceptual Reasoning, Working Memory and Processing Speed. The full version of the WISC-IV has 15 subtests, only ten are considered core, and used more often when testing intelligence.
Change from baseline Conners' Continuous Performance Test 3rd Edition (Conners CPT 3) at 14 weks | This test was administered at baseline and at week 14
  This test is a task-oriented computerized assessment of attention-related problems in individuals aged 8 years and older. By indexing the respondent's performance in areas of inattentiveness, impulsivity, sustained attention and vigilance.

OTHER OUTCOMES:
Change from baseline Conners Rating Scales Revised at 14 weeks. | This scale was administered at baseline and at week 14
  In this study we used the short parents' version (27 items) and teachers' version (28 items). The scale is divided into 4 subscales: oppositional, inattention, hyperactivity -impulsivity and ADHD Index. Each item is scored from 0 to 3 (0= not true, 3= is always true). A typical score ≥70 indicates the presence of alterations in the subscale.

CONTACTS AND LOCATIONS:
Overall Officials: M. Dolores Rodrigo Claverol, PhD, Principal Investigator — Institut Català de la Salut
Locations (2):
- Spain (2):
  - Centre Atenció Primària Bordeta-Magraners, Lleida
  - Salut Mental Infanto-Juvenil Sant Joan de Déu Terres de Lleida, Lleida